CLINICAL TRIAL: NCT01930409
Title: A Feasibility Study Investigating Telephone Supported Discharge From Acute Care to the Community After Hip Fracture
Brief Title: Back to the Future: Bridging the Hospital to Home Continuum After Hip Fracture
Acronym: B2F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Dolores Langford, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H13-01810
Record Dates: First submitted 2013-07-31; First posted 2013-08-28 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Hip Fracture
Keywords: Femoral Fractures; Hip Fractures; Frail older adults; Quality of Life; Feasibility Studies
MeSH Terms: conditions — Hip Fractures; Femoral Fractures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education Only (Active Comparator): * A 1 hour education session in the acute setting
  * A toolkit with education, exercise and self management instructions for after hip fracture
  Interventions: Behavioral: Education Only
- Education + Telephone Follow-up (Experimental): * A 1 hour education session in the acute setting
  * A telephone delivered self management program , including a toolkit (education, exercise and self management instructions for after hip fracture), support to take an active role in recovery, including setting and monitoring goals, problem solving mobility barriers, and guidance on the recovery process following a hip fracture.
  Interventions: Behavioral: Telephone Support and Coaching; Behavioral: Education Only

INTERVENTIONS:
Behavioral: Telephone Support and Coaching — The participants will receive up to 5 telephone calls of 30-45 minutes each after hospital discharge to provide support and education for the transition from acute to community care. The first call will be made within 48-72 hours of hospital discharge and will have the following elements:
  * Health Status
  * Medication Management
  * Activity/Exercise Prescription and Goal-Setting
  * Falls Prevention
  * Clarification of Appointments
  * Coordination of Post-Discharge Home Services
  * What To Do If a Problem Arises
  Arms: Education + Telephone Follow-up
Behavioral: Education Only — An educational toolkit will be provided, with materials to self manage at home after hospital discharge following a fall related hip fracture

SUMMARY:
The purpose of this study is to determine whether is is feasible and acceptable to deliver a telephone based coaching intervention compared with education alone in community dwelling older adults (age 60 and older) after a fall related hip fracture.

DETAILED DESCRIPTION:
The investigators propose a randomized controlled trial design to inform the development of a larger scale study to test effectiveness of a clinician supported telephonic self management intervention for older adults after hip fracture. The primary aim is to determine feasibility and acceptability of the intervention, and the secondary aim is to measure statistical trends on quality of life at 4 months after fracture in community dwelling older adults. In parallel, we will conduct a process evaluation to ascertain key features of the intervention via qualitative interviews of participants and health care professionals involved in delivery of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults (men and women) over 60 years of age
* Fall related hip fracture
* Community dwelling
* English speaking

Exclusion Criteria:

* Dementia
* Medical co-morbidities precluding physical activity (significant heart failure, palliative conditions etc.)
* Profound hearing loss

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of study recruitment and retention | 1 year
  Feasibility will be measured by recruitment rate (30%), and retention rate (<10% attrition)

SECONDARY OUTCOMES:
Quality of Life EQ5D-5L | 4 months
  The EQ5D-5L Quality of Life outcome measure is a self reported questionnaire measure, and has been extensively investigated in the hip fracture population, with well established sensitivity, reliability and validity properties.

OTHER OUTCOMES:
Quality of Life ICECAP-O | 4 months
de Morton Mobility Index (DEMMI) | 4 months
  The DEMMI is a clinical instrument for measuring mobility in older adults. Interval levels are obtained from 0 (poor mobility) to 100 (excellent mobility)
Gait (Walking) speed | 4 months
  Gait speed is a reliable, valid and sensitive measure likened to a vital sign.
Falls FES-1 | 4 months
  Falls self efficacy questionnaire will be used.
Pain: Visual Analogue Scale (VAS) | 4 months
Falls self report diary | 4 months
  Participants will record Falls in a check box format daily
The Hospital Anxiety and Depression Scale (HADS) | 4 months
  The HADS is a 14 item self reported questionnaire designed to assess anxiety and depression

CONTACTS AND LOCATIONS:
Overall Officials: Dolores P Langford, Msc., Principal Investigator — Vancouver Coastal Health; Maureen C Ashe, PhD, Study Director — Centre for Hip Health and Mobility
Locations (1):
- Lions Gate Hospital, North Vancouver, British Columbia, Canada